CLINICAL TRIAL: NCT00594386
Title: An Open-Label Extension to the Double-Blind SP650 Trial to Assess the Safety of Long-Term Treatment of Rotigotine in Subjects With Advanced-Stage Idiopathic Parkinson's Disease.
Brief Title: An Open-Label Extension Trial to Assess the Safety of Long-Term Treatment of Rotigotine in Advance-Stage Parkinson's Disease
Acronym: SP715
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0715
Record Dates: First submitted 2007-12-24; First posted 2008-01-15 (Estimated); Results first posted 2009-12-18 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2010-09

CONDITIONS: Parkinson's Disease
Keywords: Rotigotine; Neupro
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental)
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Rotigotine transdermal patches:
  10 cm2 (2 mg/24 hours); 20 cm2 (4 mg/24 hours); 30 cm2 (6 mg/24 hours); 40 cm2 (8 mg/24 hours)
  Optimal dosing:
  During the first year: The maximum Rotigotine dose allowed is 6 mg/24 hours.
  After the first year: Allowed dose increase of Rotigotine up to a maximum of 16 mg/24 hours.
  Other Names: Neupro

SUMMARY:
The objective of this open-label extension is to assess the safety and tolerability of long-term treatment of the Rotigotine patch in subjects with advanced-stage idiopathic Parkinson's Disease.

DETAILED DESCRIPTION:
This is the open-label extension to the randomized, double-blind, placebo-controlled SP650 trial that assessed the efficacy and safety and tolerability of the Rotigotine patch in subjects with advanced-stage idiopathic Parkinson's Disease who are not well-controlled on Levodopa.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed six months of maintenance treatment in the SP650 double-blind trial

Exclusion Criteria:

* Subjects who had an ongoing serious adverse event from the SP650 double-blind trial that was assessed as related to study medication

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2002-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (41):
- United States (37):
  - Huntsville, Alabama
  - Peoria, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Fountain Valley, California
  - Fresno, California
  - Irvine, California
  - Los Angeles, California
  - Danbury, Connecticut
  - Fairfield, Connecticut
  - New Haven, Connecticut
  - Miami, Florida
  - Pompano Beach, Florida
  - St. Petersburg, Florida
  - Sunrise, Florida
  - Atlanta, Georgia
  - Hoffman Estates, Illinois
  - Fort Wayne, Indiana
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - Henderson, Nevada
  - Albany, New York
  - Forest Hills, New York
  - Louisville, New York
  - Asheville, North Carolina
  - Raleigh, North Carolina
  - Toledo, Ohio
  - Upland, Pennsylvania
  - Houston, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Roanoke, Virginia
  - Milwaukee, Wisconsin
- Canada (4):
  - Edmonton, Alberta
  - Ottawa, Ontario
  - Montrél, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multicenter Open-Label Extension Trial to Assess the Safety of Long-Term Treatment of Rotigotine in Advanced-Stage Parkinson's Disease with 41 sites in United States and Canada from August 2002 to December 2008
Groups:
- Rotigotine: Optimal dosing for Rotigotine transdermal patches, once daily: Year 1, the maximum dose allowed is 6 mg/24 hours. After Year 1, a dose increase is allowed up to a maximum of 16 mg/24 hours.
Period: Overall Study
Arm/Group | Rotigotine
Started | 258
Completed | 0 (Study fully recruited. Completed upon market authorization and commercial availability of Neupro.)
Not Completed | 258
Not completed — Major protocol violation | 2
Not completed — Lack of Efficacy | 12
Not completed — Adverse Event | 68
Not completed — Unsatisfactory compliance of subject | 11
Not completed — Subject withdrew consent | 35
Not completed — Study ended per sponsor | 115
Not completed — Lost to Follow-up | 6
Not completed — Other: Patient went off patch (hospital) | 1
Not completed — Other: Subject moved to Seattle | 1
Not completed — Other: Subject admitted to nursing home | 1
Not completed — Other: Study terminated per investigator | 2
Not completed — Other: Sponsor closure of study | 1
Not completed — Other: Site terminated participation | 1
Not completed — Other: Patient wants prescription Neupro | 1
Not completed — Other: Loss of drivers license | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rotigotine
Number analyzed (Participants) | 258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 98
  >=65 years | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 173
Region of Enrollment [Number; unit: participants]
  United States | 243
  Canada | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Adverse Event During This Open-label Extension Study
Description: Adverse events are any untoward medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: 6 years
Population: Of the 258 subjects who entered the study, 258 are included in this summary based on the Safety Set (SS).
Measure: Number; unit: Subjects
Arm/Group | Rotigotine
Number analyzed (Participants) | 258
Subjects | 258

2. Secondary Outcome: Number of Subjects Who Withdrew From the Trial Due to an Adverse Event.
Description: as for outcome 1
Time Frame: 6 years
Population: Of the 258 subjects who entered the study, 258 are included in this summary based on the Safety Set (SS).
Measure: Number; unit: Subjects
Arm/Group | Rotigotine
Number analyzed (Participants) | 258
Subjects | 68

3. Secondary Outcome: Mean Epworth Sleepiness Scale Score During the Open-label Extension.
Description: The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. The total ESS score is the sum of 8 item-scores and can range between 0 and 24. The higher the score, the higher the person's level of daytime sleepiness.
Time Frame: Visit 11 (end of year 1), Visit 15 (end of year 2), Visit 19 (end of year 3), Visit 23 (end of year 4), Visit 27 (end of year 5), Visit 31 (end of year 6), End of Treatment (last study visit or early withdrawal visit)
Population: Of the 258 subjects who entered the study, 258 are included in this summary based on the Safety Set (SS). Last observation carried forward (LOCF) was utilized.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 258
Score on a scale
  Visit 11 (end of year 1) (n=254) | 8.6 (4.9)
  Visit 15 (end of year 2) (n=254) | 8.9 (4.9)
  Visit 19 (end of year 3) (n=254) | 9.3 (5.1)
  Visit 23 (end of year 4) (n=254) | 9.8 (5.2)
  Visit 27 (end of year 5) (n=254) | 9.7 (5.3)
  Visit 31 (end of year 6) (n=254) | 10.0 (5.4)
  End of Treatment (n=258) | 10.0 (5.4)

ADVERSE EVENTS:
Time Frame: Up to 6 years
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 165/258
Other Adverse Events (participants affected / at risk) | 253/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=258)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 5 (5)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (2)
Angina unstable (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 7 (12)
Coronary artery disease (Cardiac disorders) | 6 (6)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Cardiac aneurysm (Cardiac disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (4)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (3)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 10 (11)
Pain (General disorders) | 1 (1)
Asthenia (General disorders) | 3 (3)
Malaise (General disorders) | 1 (1)
Implant site pain (General disorders) | 1 (1)
Mechanical complication of implant (General disorders) | 1 (1)
Implant site erosion (General disorders) | 1 (1)
Gait disturbance (General disorders) | 2 (2)
Cardiac death (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 6 (8)
Bronchitis (Infections and infestations) | 3 (3)
Lobar pneumonia (Infections and infestations) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Bronchitis acute (Infections and infestations) | 1 (2)
Cellulitis (Infections and infestations) | 7 (8)
Arthritis bacterial (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (9)
Device related infection (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Incision site abscess (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Rectal abscess (Infections and infestations) | 1 (1)
Extradural abscess (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Cellulitis streptococcal (Infections and infestations) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 13 (14)
Hip fracture (Injury, poisoning and procedural complications) | 6 (6)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 5 (5)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2)
Hepatic trauma (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (4)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (2)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 9 (9)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Parkinson's disease (Nervous system disorders) | 25 (28)
Parkinsonian crisis (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 8 (9)
Embolic stroke (Nervous system disorders) | 2 (2)
Brain stem infarction (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 8 (9)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 4 (5)
Dyskinesia (Nervous system disorders) | 3 (3)
Akinesia (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 8 (8)
Hallucination, visual (Psychiatric disorders) | 2 (2)
Mental status changes (Psychiatric disorders) | 3 (3)
Confusional state (Psychiatric disorders) | 3 (3)
Sleep attacks (Psychiatric disorders) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Pathological gambling (Psychiatric disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (3)
Acute prerenal failure (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Nephrosclerosis (Renal and urinary disorders) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep brain stimulation (Surgical and medical procedures) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 2 (3)
Haemorrhage (Vascular disorders) | 2 (2)
Circulatory collapse (Vascular disorders) | 2 (2)
Aortic stenosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (2)
Arteriosclerosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=258)
Anaemia (Blood and lymphatic system disorders) | 18 (19)
Cataract (Eye disorders) | 24 (33)
Constipation (Gastrointestinal disorders) | 58 (66)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 (23)
Nausea (Gastrointestinal disorders) | 61 (94)
Vomiting (Gastrointestinal disorders) | 29 (32)
Diarrhoea (Gastrointestinal disorders) | 25 (28)
Abdominal pain (Gastrointestinal disorders) | 13 (17)
Dyspepsia (Gastrointestinal disorders) | 13 (14)
Application site erythema (General disorders) | 37 (44)
Application site pruritus (General disorders) | 34 (35)
Application site reaction (General disorders) | 14 (16)
Oedema peripheral (General disorders) | 80 (111)
Fatigue (General disorders) | 22 (23)
Asthenia (General disorders) | 18 (20)
Upper respiratory tract infection (Infections and infestations) | 39 (51)
Nasopharyngitis (Infections and infestations) | 32 (41)
Urinary tract infection (Infections and infestations) | 55 (86)
Pneumonia (Infections and infestations) | 14 (15)
Cellulitis (Infections and infestations) | 18 (21)
Fall (Injury, poisoning and procedural complications) | 100 (198)
Excoriation (Injury, poisoning and procedural complications) | 17 (26)
Contusion (Injury, poisoning and procedural complications) | 29 (54)
Skin laceration (Injury, poisoning and procedural complications) | 23 (30)
Weight decreased (Investigations) | 24 (26)
Dehydration (Metabolism and nutrition disorders) | 15 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 51 (65)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 46 (65)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 35 (46)
Neck pain (Musculoskeletal and connective tissue disorders) | 17 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 60 (77)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 24 (30)
Arthritis (Musculoskeletal and connective tissue disorders) | 17 (18)
Somnolence (Nervous system disorders) | 150 (236)
Dizziness (Nervous system disorders) | 61 (72)
Hypoaesthesia (Nervous system disorders) | 20 (25)
Parkinson's disease (Nervous system disorders) | 20 (22)
Headache (Nervous system disorders) | 28 (36)
Dyskinesia (Nervous system disorders) | 25 (32)
Memory impairment (Nervous system disorders) | 15 (15)
Balance disorder (Nervous system disorders) | 13 (13)
Hallucination (Psychiatric disorders) | 54 (68)
Insomnia (Psychiatric disorders) | 56 (66)
Depression (Psychiatric disorders) | 46 (51)
Confusional state (Psychiatric disorders) | 39 (44)
Anxiety (Psychiatric disorders) | 34 (38)
Urinary incontinence (Renal and urinary disorders) | 28 (30)
Pollakiuria (Renal and urinary disorders) | 17 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (30)
Rash (Skin and subcutaneous tissue disorders) | 23 (26)
Hypertension (Vascular disorders) | 36 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.